CLINICAL TRIAL: NCT03015116
Title: Effectiveness of Photobiomodulation Compared to Usual Care for Plantar Fasciitis
Brief Title: Photobiomodulation for Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Landstuhl Regional Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ann Ketz, Chief, Center for Nursing Science and Clinical Inquiry, Landstuhl Regional Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M-10548
Record Dates: First submitted 2017-01-04; First posted 2017-01-09 (Estimated); Results first posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Plantar Fascitis
Keywords: photobiomodulation; plantar fasciitis
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Cryotherapy; Ice; Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Care (Active Comparator): Participants will complete 6 weeks of stretching and cryotherapy
  Interventions: Other: Stretching; Other: Cryotherapy
- PBM 10 Watts (Experimental): Participants will complete 6 weeks of stretching and cryotherapy, plus 9 treatments of PBM (810/980 nm continuous wave, 10 Watts power) over 3 weeks
  Interventions: Other: Stretching; Other: Cryotherapy; Device: Photobiomodulation Low Power
- PBM 25 Watts (Experimental): Participants will complete 6 weeks of stretching and cryotherapy, plus 9 treatments of PBM (810/980 nm continuous wave, 25 Watts power) over 3 weeks
  Interventions: Other: Stretching; Other: Cryotherapy; Device: Photobiomodulation High Power

INTERVENTIONS:
Other: Stretching — Daily foot and ankle stretching protocol
Other: Cryotherapy — Daily cryotherapy in conjunction with stretching
  Other Names: Ice
Device: Photobiomodulation Low Power — Photobiomodulation treatment with 10W power output
  Other Names: Low Level Laser therapy; low level light therapy
  Arms: PBM 10 Watts
Device: Photobiomodulation High Power — Photobiomodulation treatment with 25W power output
  Other Names: Low level laser therapy; low level light therapy
  Arms: PBM 25 Watts

SUMMARY:
BACKGROUND: Plantar fasciitis, a degenerative injury of the connective tissue in the foot, results in pain-related disability in Service Members and beneficiaries and contributes to decreased physical activity and excessive healthcare costs. Even if effective, current treatment protocols may require 6-12 months of therapy to return individuals to pain-free activity. Photobiomodulation (PBM), or low level laser therapy, uses non-ionizing light to elicit biological changes in tissues resulting in beneficial therapeutic outcomes. Evidence supports use of PBM for other degenerative connective tissue conditions, such as Achilles tendinopathy and epicondylitis. Unfortunately, previous studies of PBM for treatment of plantar fasciitis lack optimized treatment parameters and therefore have been inconclusive on its clinical effectiveness.

SPECIFIC AIMS: 1. Establish feasibility of and adherence to a photobiomodulation protocol in conjunction with and compared to usual care for plantar fasciitis treatment. 2. Assess the clinical effectiveness of photobiomodulation in conjunction with and compared to usual care to improve function and decrease pain and in patients. 3. Assess the difference between two photobiomodulation dose parameters in conjunction with and compared to usual care for plantar fasciitis treatment.

DESIGN: The investigators will use a prospective randomized controlled trial to meet the aims of this exploratory study. METHOD: A sample of 114 military healthcare beneficiaries will be randomly assigned to either usual care, usual care plus PBM lower dose, or usual care plus PBM higher dose groups. At baseline, during the treatment protocol, and at long term (3 and 6 month) follow-up, measures of foot function and pain will be collected for analysis. The proposed methods will allow the study team to establish if PBM accelerates recovery compared to usual care, as well as determining the optimal dose for future trials comparing PBM to other, more invasive, therapies for plantar fasciitis.

ELIGIBILITY:
Inclusion Criteria:

1. Between ages of 18 - 65 years
2. Eligible for care at Landstuhl Regional Medical Center
3. Diagnosis of PF by healthcare provider based on accepted diagnostic criteria
4. Have experienced symptoms of PF for at least 3 months
5. Able to read and understand English language for consent purposes
6. Able to commit to 6 week intervention and 3 and 6 month follow-up

Exclusion Criteria:

1. Pregnant or plan on becoming pregnant during intervention period (Safety of PBM not established in pregnancy)
2. History of traumatic injury to symptomatic foot/feet
3. Diagnosis of calcaneal fracture
4. Have previously had corticosteroid injections, surgery, or other invasive treatment for same condition
5. Greater than 15% of calf area covered in tattoos/ink/scarring (Pigment in ink can absorb light, causing overheating of skin)
6. History of neuropathy or unable to detect changes in skin temperature (increased risk of skin warming due to inability to detect change)
7. Currently using medications associated with sensitivity to heat or light (e.g. amiodarone, chlorpromazine, doxycycline, hydrochlorothiazide, nalidixic acid, naproxen, piroxicam, tetracycline, thioridazine, voriconazole)(8) Concurrent participation in another research study addressing pain issue

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann K Ketz, PhD, Principal Investigator — LRMC
Locations (1):
- Landstuhl Regional Medical Center, Landstuhl, APO AE, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | PBM 10 Watts | PBM 25 Watts
Started | 38 | 38 | 38
Completed | 31 | 36 | 36
Not Completed | 7 | 2 | 2
Not completed — Lost to Follow-up | 3 | 0 | 2
Not completed — Withdrawal by Subject | 3 | 1 | 0
Not completed — Subject has New Medical Status | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | PBM 10 Watts | PBM 25 Watts | Total
Number analyzed (Participants) | 38 | 38 | 38 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 37 | 38 | 38 | 113
  >=65 years | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 25 | 22 | 64
  Male | 21 | 13 | 16 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 23 | 21 | 23 | 67
  African-American | 6 | 6 | 7 | 19
  Hispanic/Latino | 4 | 4 | 5 | 13
  American Indian | 0 | 1 | 0 | 1
  Asian/Pacific Islander | 4 | 2 | 3 | 9
  Other | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Germany | 38 | 38 | 38 | 114
Body Mass Index [Count of Participants; unit: Participants]
  Underweight (Less than 18.5) | 0 | 0 | 1 | 1
  Normal Weight (18.5 - 24.9) | 3 | 7 | 4 | 14
  Overweight (25-29.9) | 18 | 23 | 16 | 57
  Obese (Greater than or Equal to 30.0) | 17 | 8 | 17 | 42
Number of Months with Plantar Fasciitis or Plantar Heel Pain [Count of Participants; unit: Participants]
  0 to 6 Months | 8 | 4 | 8 | 20
  7 to 12 Months | 10 | 7 | 6 | 23
  13 to 24 Months | 6 | 5 | 8 | 19
  Greater than 24 months | 14 | 18 | 16 | 48
  Missing Data | 0 | 4 | 0 | 4
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — A numerical schema for skin color based on melanin pigment, which participants self-select. There is no inherent value to the numbers. 1- skin ivory, always freckles, always burns/peels, never tans; 2 - skin fair or pale, usually freckles, burns/peels often, rarely tans; 3 - skin fair to beige, might freckle, burns on occasion, sometimes tans; 4 - skin olive or light brown, doesn't really freckle, burns rarely, tans often; 5 - skin dark brown, rarely freckles, almost never burns, always tans; 6 - skin deeply pigmented dark brown, never freckles, never burns, always tans darkly.
  Participants
    Type I | 1 | 2 | 2 | 5
    Type II | 7 | 5 | 2 | 14
    Type III | 14 | 17 | 13 | 44
    Type IV | 8 | 8 | 13 | 29
    Type V | 7 | 5 | 7 | 19
    Type VI | 0 | 1 | 1 | 2
    Missing Data | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Foot and Ankle Ability Measure (FAAM)
Description: The FAAM is a 29-item self-report instrument that assesses physical function in foot and ankle impairments which included plantar fasciitis cases in development. There are two subscales, Activities of Daily Living (21-item) and Sports (8-item). Each item is scored on a 5-point Likert scale (4='no difficulty at all' to 0='unable to do'); points are transformed to a percentage (100%=no dysfunction). A higher score means a better outcome.
Time Frame: Baseline, 3 weeks, and 6 weeks
Population: 7 withdrew from Usual Care group; 2 each from treatment groups.
Measure: Mean (95% Confidence Interval); unit: percentage of total score
Arm/Group | Usual Care | PBM 10 Watts | PBM 25 Watts
Number analyzed (Participants) | 31 | 36 | 36
percentage of total score
  Baseline ADL Subscale | 66.2 [61.2 to 71.2] | 72.4 [67.3 to 77.4] | 69.9 [64.8 to 74.9]
  Week 3 ADL Subscale | 69.3 [63.9 to 74.9] | 81.4 [76.2 to 86.5] | 78.5 [73.4 to 83.6]
  Week 6 ADL Subscale | 70.4 [65.1 to 75.7] | 82.9 [77.7 to 88.0] | 82.3 [77.2 to 87.4]
  Baseline Sports Subscale | 46.4 [39.4 to 53.3] | 46.5 [39.5 to 53.5] | 46.3 [39.3 to 53.3]
  Week 3 Sports Subscale | 46.6 [39.2 to 54.0] | 62.4 [55.3 to 69.5] | 62.0 [55.1 to 68.9]
  Week 6 Sports Subscale | 53.9 [46.6 to 61.1] | 67.7 [60.6 to 74.4] | 65.7 [58.7 to 72.7]

2. Primary Outcome: Defense and Veterans Pain Rating Scale (DVPRS)
Description: Defense and Veterans Pain Rating Scale (DVPRS). This 5-item scale integrates a numeric pain rating scale with visual facial cues and word descriptors as well as 4 supplemental questions on pain interference. Each item is scores 0-10 with higher scores indicating worse pain/interference. Lower scores mean a better outcome.
Time Frame: Baseline, 3 weeks, and 6 weeks
Population: 7 withdrew from Usual Care group; 2 each from treatment groups.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Usual Care | PBM 10 Watts | PBM 25 Watts
Number analyzed (Participants) | 31 | 36 | 36
score on a scale
  Baseline 24 Hour Pain | 4.031 [3.215 to 4.848] | 4.146 [3.505 to 4.786] | 3.763 [3.110 to 4.415]
  Week 3 24 Hour Pain | 3.634 [2.658 to 4.610] | 2.948 [2.182 to 3.714] | 2.863 [2.082 to 3.644]
  Week 6 24 Hour Pain | 3.652 [2.695 to 6.608] | 2.61 [1.859 to 3.360] | 2.943 [2.178 to 3.708]
  Baseline Activity Interference | 3.462 [2.516 to 4.408] | 3.869 [3.169 to 4.570] | 3.798 [3.018 to 4.578]
  Week 3 Activity Interference | 3.513 [2.522 to 4.503] | 2.696 [1.962 to 3.430] | 2.777 [1.960 to 3.594]
  Week 6 Activity Interferece | 3.555 [2.608 to 4.501] | 2.244 [1.543 to 2.945] | 2.736 [1.955 to 3.516]
  Baseline Sleep Interference | 1.857 [0.966 to 2.748] | 2.548 [1.888 to 3.207] | 1.667 [0.932 to 2.401]
  Week 3 Sleep Interference | 2.269 [1.336 to 3.202] | 1.986 [1.296 to 2.677] | 1.229 [0.460 to 1.998]
  Week 6 Sleep Interference | 1.748 [0.900 to 2.596] | 1.476 [0.848 to 2.104] | 1.111 [0.412 to 1.811]
  Baseline Mood Interference | 2.496 [1.577 to 3.414] | 2.363 [1.682 to 3.043] | 2.164 [1.406 to 2.921]
  Week 3 Mood Interference | 2.630 [1.662 to 3.599] | 1.530 [0.813 to 2.247] | 1.589 [0.790 to 2.387]
  Week 6 Mood Interference | 2.092 [1.212 to 2.973] | 1.125 [0.473 to 1.777] | 1.486 [0.760 to 2.211]
  Baseline Stress Interference | 2.471 [1.489 to 3.462] | 2.358 [1.631 to 3.085] | 2.215 [1.406 to 3.024]
  Week 3 Stress Interference | 2.504 [1.534 to 3.475] | 1.433 [0.770 to 2.207] | 1.646 [0.846 to 2.446]
  Week 6 Stress Interference | 2.345 [1.441 to 3.248] | 1.031 [0.62 to 1.699] | 1.450 [0.705 to 2.195]

3. Primary Outcome: Foot and Ankle Ability Measure (FAAM) Long-term
Description: as for outcome 1
Time Frame: 3 months and 6 months
Population: Individuals were lost to follow up at each long term follow up time point. Participants from the UC group completed the study after the 6 week follow-up time point. No data were collected from UC care group for the 3 and 6 month time points, therefore are not included in the 3 and 6 month measures.
Measure: Mean (95% Confidence Interval); unit: percentage of total score
Arm/Group | PBM 10 Watts | PBM 25 Watts
Number analyzed (Participants) | 28 | 36
percentage of total score
  3 Months ADL Subscale | 80.3 [74.6 to 85.9] | 81.5 [76.1 to 86.8]
  3 Months Sports Subscale | 62.4 [53.9 to 70.9] | 67.6 [59.6 to 75.7]
  6 Months ADL Subscale: number analyzed (Participants) | 25 | 30
  6 Months ADL Subscale | 82.0 [76.1 to 87.9] | 82.2 [76.7 to 87.8]
  6 Months Sports Subscale: number analyzed (Participants) | 25 | 30
  6 Months Sports Subscale | 65.4 [56.5 to 74.3] | 69.0 [60.6 to 77.3]

4. Primary Outcome: Defense and Veterans Pain Rating Scale (DVPRS) Long-term
Description: as for outcome 2
Time Frame: 3 months and 6 months
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PBM 10 Watts | PBM 25 Watts
Number analyzed (Participants) | 28 | 36
score on a scale
  Month 3 24 Hour Pain | 2.449 [1.688 to 3.211] | 1.977 [1.315 to 2.639]
  Month 6 24 Hour Pain: number analyzed (Participants) | 25 | 30
  Month 6 24 Hour Pain | 2.126 [1.350 to 2.901] | 2.148 [1.450 to 2.847]
  Month 3 Activity Interference | 2.583 [1.828 to 3.337] | 1.995 [1.286 to 2.704]
  Month 6 Activity Interference: number analyzed (Participants) | 25 | 30
  Month 6 Activity Interference | 2.326 [1.540 to 3.113] | 1.818 [1.094 to 2.542]
  Month 3 Sleep Interference | 1.691 [0.974 to 2.409] | 0.720 [0.146 to 1.294]
  Month 6 Sleep Interference: number analyzed (Participants) | 25 | 30
  Month 6 Sleep Interference | 1.541 [0.796 to 2.287] | 0.880 [0.149 to 1.294]
  Month 3 Mood Interference | 1.770 [1.094 to 2.445] | 1.034 [0.399 to 1.669]
  Month 6 Mood Interference: number analyzed (Participants) | 25 | 30
  Month 6 Mood Interference | 1.614 [0.910 to 2.317] | 1.157 [0.509 to 1.805]
  Month 3 Stress Interference | 1.174 [0.484 to 1.864] | 1.040 [0.378 to 1.702]
  Month 6 Stress Interference: number analyzed (Participants) | 25 | 30
  Month 6 Stress Interference | 1.391 [0.579 to 2.204] | 1.040 [0.261 to 1.819]

5. Secondary Outcome: Ankle Dorsiflexion
Description: Measures range of motion of ankle in weight-bearing conditions; recorded as distance from great toe to wall at maximal dorsiflexion in centimeters. The percentage of change between timepoints will be calculated for each individual and then compiled per group.
Time Frame: % change from baseline to 3 weeks, % change from 3 weeks to 6 weeks, % change from baseline to 6 weeks
Measure: Mean (Standard Error); unit: percentage of change over time
Arm/Group | Usual Care | PBM 10 Watts | PBM 25 Watts
Number analyzed (Participants) | 30 | 35 | 35
percentage of change over time
  % Change baseline to 3 weeks | 9.14 (0.029) | 7.16 (0.036) | 17.24 (0.045)
  % change week 3 to week 6 | 6.03 (0.037) | 9.02 (0.047) | 3.86 (0.023)
  % change baseline to week 6 | 11.6 (0.055) | 13.22 (0.043) | 19.79 (0.045)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the six weeks of active study treatment.
Arm/Group | Usual Care | PBM 10 Watts | PBM 25 Watts
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 0/38 | 1/38 | 0/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=38) | PBM 10 Watts (N=38) | PBM 25 Watts (N=38)
Numbness and Tingling (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Grade 2, probably not related to treatment

LIMITATIONS AND CAVEATS:
No sham group to neutralize bias related to intervention; Not able to compare the usual care group to the intervention group in long term follow up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT03015116/Prot_SAP_000.pdf
  • Informed Consent Form (2016-11-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT03015116/ICF_001.pdf